CLINICAL TRIAL: NCT00170768
Title: Cognitive Effects of Darifenacin and Oxybutynin Extended Release in Volunteers Aged 60 and Over
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDAR328A2403
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Healthy Volunteers
Keywords: Darifenacin, oxybutynin, cognition, memory
MeSH Terms: interventions — darifenacin; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Active Comparator): Oxybutynin
  Interventions: Drug: Oxybutynin
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin — Darifenacin modified release 7,5 mg tablets once daily titrated to 15 mg once daily
  Other Names: Enablex
  Arms: 1
Drug: Oxybutynin — Oxybutynin extended release 10 mg tablet once daily titrated to 15 mg, then to 20 mg once daily
  Arms: 2
Drug: Placebo — Placebo once daily tablet (sham titration)
  Arms: 3

SUMMARY:
The purpose of this study is to explore the possible cognitive effects of darifenacin modified release and long-acting oxybutynin.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 60 and over
* United States English as a primary language
* Given written informed consent by signing and dating an informed consent form prior to study entry

Exclusion Criteria:

* Current diseases in which the use of anti-cholinergic drugs is contraindicated, including the use of drugs with anti-cholinergic effects
* Volunteers with history of urinary retention or current bladder outlet obstruction, as determined by the investigator

Other protocol defined inclusion/exclusion criteria may apply.

- Current use of drugs known to effect memory and cognition Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-02; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Cognitive effect: measure of accuracy of delayed recall name-phase association test at week 3.

SECONDARY OUTCOMES:
Cognitive effect: measure of accuracy of delayed recall name-phase association test at week 1 & 2.
Effects on other cognitive domains measured by various tests at week 1,2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Washington Neuropsychological Institute LLC Georgetown, Washington D.C., District of Columbia, United States